CLINICAL TRIAL: NCT01412034
Title: Modifying Orphan Disease Evaluation (MODE) Study: A Multicenter, Open-label Study of the Effects of CER-001 on Plaque Volume in Subjects With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: Effect of CER-001 on Plaque Volume in Homozygous Familial Hypercholesterolemia (HoFH) Subjects
Acronym: MODE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerenis Therapeutics, SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER-001-CLIN-003
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: Homozygous Familial Hypercholesterolemia; Familial Hypercholesterolemia; HDL mimetic; ApoA-1
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — CER-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CER-001 (Experimental): Open label single arm study of CER-001
  Interventions: Drug: CER-001

INTERVENTIONS:
Drug: CER-001 — Biweekly infusion

SUMMARY:
The available medications used to treat HoFH are targeted at reducing circulating levels of total and LDL-cholesterol. These measures can retard the progression of cardiovascular disease, however, they are unlikely to regress existing disease due to years of cholesterol accumulation in the vessel walls and therefore cannot adequately reduce the existing risk for an ischemic event. HDL has multiple actions that could lead to plaque stabilization and regression, such as rapid removal of large quantities of cholesterol from the vasculature, improvement in endothelial function, protection against oxidative damage and reduction in inflammation. This study will assess the effects of CER-001, a recombinant human Apo-A-1 based HDL mimetic, on indices of atherosclerotic plaque progression and regression as assessed by 3Tesla MRI measurements in patients with HoFH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 12 years or older
* Subject presents with Homozygous FH

Exclusion Criteria:

* Weight >100 kg
* Subjects with significant health problems in the recent past including blood disorders, cancer, or digestive problems
* Female subjects of child-bearing potential
* Known major hematologic, renal , hepatic, metabolic, gastrointestinal or endocrine dysfunction
* Contraindication to MRI scanning that would preclude the use of contrast-enhanced 3TMRI

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to follow-up in carotid mean vessel wall area | Baseline then 6 months and/or ~2 weeks post final dose
  Percent change from baseline to follow-up in carotid mean vessel wall area

SECONDARY OUTCOMES:
Change in carotid vessel wall volume | Baseline then 6 months and/or ~2 weeks post final dose
  Percent change in carotid vessel wall volume , as assessed by 3TMRI, from the baseline measurement to the follow up taken ~2 weeks following the final dose of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: John J. Kastelein, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (9):
- United States (2):
  - Clinical Research Facility, Hartford, Connecticut
  - Clinical Research Facility, North Massapequa, New York
- Canada (2):
  - Clinical Research Facility, Chicoutimi, Quebec
  - Clinical Research Facility, Québec, Quebec
- Clinical Research Facility, Rome, Italy
- Netherlands (3):
  - Clinical Research Facility, Amsterdam
  - Clinical Research Facility, Maastricht
  - Clinical Research Facility, Nijmegen
- Clinical Research Facility, Manchester, United Kingdom

REFERENCES:
- [Background] Eriksson M, Carlson LA, Miettinen TA, Angelin B. Stimulation of fecal steroid excretion after infusion of recombinant proapolipoprotein A-I. Potential reverse cholesterol transport in humans. Circulation. 1999 Aug 10;100(6):594-8. doi: 10.1161/01.cir.100.6.594. PMID 10441095
- [Background] Nanjee MN, Doran JE, Lerch PG, Miller NE. Acute effects of intravenous infusion of ApoA1/phosphatidylcholine discs on plasma lipoproteins in humans. Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):979-89. doi: 10.1161/01.atv.19.4.979. PMID 10195926
- [Background] Nieuwdorp M, Vergeer M, Bisoendial RJ, op 't Roodt J, Levels H, Birjmohun RS, Kuivenhoven JA, Basser R, Rabelink TJ, Kastelein JJ, Stroes ES. Reconstituted HDL infusion restores endothelial function in patients with type 2 diabetes mellitus. Diabetologia. 2008 Jun;51(6):1081-4. doi: 10.1007/s00125-008-0975-2. Epub 2008 Apr 4. No abstract available. PMID 18389214
- [Background] Shaw JA, Bobik A, Murphy A, Kanellakis P, Blombery P, Mukhamedova N, Woollard K, Lyon S, Sviridov D, Dart AM. Infusion of reconstituted high-density lipoprotein leads to acute changes in human atherosclerotic plaque. Circ Res. 2008 Nov 7;103(10):1084-91. doi: 10.1161/CIRCRESAHA.108.182063. Epub 2008 Oct 2. PMID 18832751
- [Background] Nissen SE, Tsunoda T, Tuzcu EM, Schoenhagen P, Cooper CJ, Yasin M, Eaton GM, Lauer MA, Sheldon WS, Grines CL, Halpern S, Crowe T, Blankenship JC, Kerensky R. Effect of recombinant ApoA-I Milano on coronary atherosclerosis in patients with acute coronary syndromes: a randomized controlled trial. JAMA. 2003 Nov 5;290(17):2292-300. doi: 10.1001/jama.290.17.2292. PMID 14600188
- [Background] Tardif JC, Gregoire J, L'Allier PL, Ibrahim R, Lesperance J, Heinonen TM, Kouz S, Berry C, Basser R, Lavoie MA, Guertin MC, Rodes-Cabau J; Effect of rHDL on Atherosclerosis-Safety and Efficacy (ERASE) Investigators. Effects of reconstituted high-density lipoprotein infusions on coronary atherosclerosis: a randomized controlled trial. JAMA. 2007 Apr 18;297(15):1675-82. doi: 10.1001/jama.297.15.jpc70004. Epub 2007 Mar 26. PMID 17387133
- [Background] Waksman R, Torguson R, Kent KM, Pichard AD, Suddath WO, Satler LF, Martin BD, Perlman TJ, Maltais JA, Weissman NJ, Fitzgerald PJ, Brewer HB Jr. A first-in-man, randomized, placebo-controlled study to evaluate the safety and feasibility of autologous delipidated high-density lipoprotein plasma infusions in patients with acute coronary syndrome. J Am Coll Cardiol. 2010 Jun 15;55(24):2727-35. doi: 10.1016/j.jacc.2009.12.067. PMID 20538165
- [Result] Spieker LE, Sudano I, Hurlimann D, Lerch PG, Lang MG, Binggeli C, Corti R, Ruschitzka F, Luscher TF, Noll G. High-density lipoprotein restores endothelial function in hypercholesterolemic men. Circulation. 2002 Mar 26;105(12):1399-402. doi: 10.1161/01.cir.0000013424.28206.8f. PMID 11914243